CLINICAL TRIAL: NCT03300739
Title: Phenotypic Measurements and Their Relation to Disease Exacerbation in COPD Patients
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ResMed (Industry)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Dermatologist, Massachusetts General Hospital
Other Study IDs: 2016P002312
Record Dates: First submitted 2017-08-23; First posted 2017-10-03 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: COPD Exacerbation; Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is an observational pilot study focused on collecting data on clinical variables that can improve the understanding of potential predictors of disease exacerbation and readmissions in COPD patients. The study aim is to understand how the variability of clinical parameters (respiratory rate, forced expiratory volume in one second, and oxygen saturation), physical activity and quality of life is associated with the risk of exacerbation in COPD patients.

DETAILED DESCRIPTION:
The investigational product to be used in this trial is the ResMed Biomotion Sensor (ResMed Sensor Technologies, Dublin, Ireland). This device uses very low power radio waves (~1/100th of the strength of a mobile phone signal) to detect respiratory movements of a person while asleep- without physical contact with the individual. The device is designed to measure up to 5 feet, so that only the person on the side of the bed nearest the device is monitored. Algorithms have been developed to analyze the respiratory movement signals and extract information about respiration rate, bodily movements, sleep/wake patterns and sleep disordered respiration.

ELIGIBILITY:
Inclusion Criteria:

1. Medically stable and ambulatory COPD (primary diagnosis) patients who have had an emergency room visit or hospitalization for an acute exacerbation of COPD within the past 30 days.
2. Sufficient understanding of the English language to be able to read and understand study procedures.

Exclusion Criteria:

1. Currently on admission in the hospital, on non-invasive positive airway pressure ventilation
2. Visual, hearing or cognitive impairments at the discretion of their physician.
3. Currently participating in a COPD telemonitoring program.
4. No AT&T cellular coverage at their primary residence
5. Any other medical or psychological condition that, in the opinion of the investigator may present an unreasonable risk to the study participant as a result of his/her participation in this study, may make participant's participation unreliable, or may interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Respiratory rate (breaths per minute) | Daily, 16 weeks
  Collected by study device, Reassure Respiration Monitor. This device uses very low power radio waves to detect respiratory movements of a person while asleep.

SECONDARY OUTCOMES:
Oxygen saturation (%) | Daily for 16 weeks
  Collected via pulse oximeter.
Forced Expiratory Volume in 1 Second (FEV1). FEV1 is the volume of air forcefully exhaled in 1 second. | Weekly for16 weeks
  Collected via spirometer
Physical activity | Daily for 16 weeks
  Collected via step counts
Body Mass Index (kg/m^2) | Baseline (Day 0) and Close-out (16 weeks)
  Weight and height will be combined to report BMI
Quality of life | Baseline (Day 0) and Close-out (16 weeks)
  Collected via SF-12 questionnaire
Depression | Monthly for 16 weeks
  Collected via PHQ-8 questionnaire
Anxiety | Baseline (Day 0) and Close-out (16 weeks)
  Collected via GAD-7 questionnaire
COPD symptom assessment | Weekly for 16 weeks
  Collected via CAT questionnaire
Functional impairment due to dyspnea | Weekly for 16 weeks
  Collected via mMRC dyspnea scale
Study device usability | Close-out (16 week)
  Collected via usability questionnaire
Medical treatment | Baseline (Day 0) and Close-out (16 weeks)
  Collected via electronic health record
Hospitalization records | Baseline (Day 0) and Close-out (16 weeks)
  Collected via electronic health record

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Agboola, MD, Principal Investigator — MGH
Locations (1):
- Partners Connected Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No